CLINICAL TRIAL: NCT05515991
Title: Assessing the Feasibility of Self-reported MeasUrement of Physical and PsychosOcial Symptoms and Response Tool in Patients on Dialysis- Pilot Study
Brief Title: Symptom Management in Patients on Dialysis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Humber River Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 22-5199; UHNKHERGePROMSUPPORTDIALYSIS (Other: University Health Network Toronto)
Record Dates: First submitted 2022-08-16; First posted 2022-08-25 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: End-stage Kidney Disease
Keywords: end-stage renal disease; hemodialysis; dialysis; chronic kidney disease; kidney failure
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SUPPORT-DIALYSIS with Access to Output Report and Information Hub (Experimental): Feasibility of SUPPORT-Dialysis at Toronto General Hospital
  Interventions: Other: SUPPORT-DIALYSIS with Access to Output Report and Information Hub
- SUPPORT-DIALYSIS Only (Experimental): Usual Treatment at Humber River Hospital
  Interventions: Other: SUPPORT-DIALYSIS Only

INTERVENTIONS:
Other: SUPPORT-DIALYSIS with Access to Output Report and Information Hub — SUPPORT-Dialysis is a symptom assessment response toolkit, consisting of a screening and response component. Participants will be screened for symptoms and distress using an electronic assessment(ePROMs). Output reports based on ePROMs scores will be provided to patients as well as the clinical care team.
  Participants at Toronto General Hospital will complete the screening every 4 weeks for 6 months, and each time the output report will be provided to both patients and the clinical team.The second, response component of the intervention is the information support and self-management hub (https://symptomcare.org). All participants and the clinical team will be given access to this website, which provides information about self-management for patients as well as management advice for healthcare professionals.
  Arms: SUPPORT-DIALYSIS with Access to Output Report and Information Hub
Other: SUPPORT-DIALYSIS Only — SUPPORT-Dialysis screening will also be implemented at Humber River Hospital, but participants and clinical team will not be receiving the output screening report or be given access to the information hub with symptom management resources.
  Arms: SUPPORT-DIALYSIS Only

SUMMARY:
This is a parallel arm, pilot study used to examine the feasibility of electronic patient reported outcome measures (ePROMs) for symptom assessment and monitoring as well as a linked self-management support and decision support information hub (https://symptomcare.org) to facilitate symptom management for patients on maintenance hemodialysis.

Two dialysis centers will be included in the study, with one center receiving SUPPORT-Dialysis (intervention arm) and the other receiving standard care (control arm).

DETAILED DESCRIPTION:
In Canada, 20,000-25,000 patients with end-stage kidney disease (ESKD) experience a range of symptoms such as chronic pain, itchiness, fatigue, anxiety, depression and sleep disturbances [1-5]. These may impact quality of life, increase mortality, decrease treatment adherence, and increased hospitalizations [6-8]. These symptoms are under-managed and under-recognized among these patients, but screening and managing symptoms using patient reported outcomes measures (PROMs) may be a useful and inexpensive solution. PROMS have previously been used successfully in cancer care [8-9], and have potential for clinical care of patients with kidney failure as well.

Electronic collection of PROMs (ePROMs) facilitates PROMs use by allowing linkage to electronic patient records [10-11] and immediate scoring and presentation of results to patients and clinicians [12-14]. ePROMs allow the use of computer adaptive testing (CAT) to personalize questions, increase the precision of measurements and reduce survey burden [15-17]. The investigators also developed a self-management support and decision support resource hub(https://symptomcare.org) to help dialysis patients and their clinical team in identifying and managing relevant physical and psychological symptoms that require further assessment and potential intervention.

Patients will complete Patient Reported Outcome Measurement Information System (PROMIS) CAT surveys on an electronic data capture system (SUPPORT-Dialysis) every four weeks during their dialysis treatment for six months. In the intervention, patients with moderate/severe symptoms will be flagged for the clinical team. Moderate/severe symptoms will be determined based on whether the participants score above a pre-defined cut-off in the surveys. The participant, primary nurse, and nephrologist will also receive an output report and be given access to https://symptomcare.org for suggested symptom management actions.

To establish the feasibility and acceptability of the intervention, the investigators will assess

1. Recruitment Rate
2. Retention and Completion rate
3. Acceptability
4. Patient satisfaction
5. Staff satisfaction

Based on the objectives of this study, the investigators hypothesize the following:

1. Recruitment goals will be met; >50% of approached patients will consent; completion rate will be > 80% of participants at least 50% of the time, and dropout rate will be < 30%.
2. >80% of patients find the toolkit acceptable; <20% of staff find the process intrusive to workflow.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing maintenance hemodialysis for more than 3 months

Exclusion Criteria:

* Patients with severe acute illness or condition that hampers questionnaire completion assessed by clinical team.
* Dementia indicated in the medical record, indicated by the managing healthcare team.
* Unable to understand English - as assessed by clinical team.
* Life expectancy < 6 months as assessed by main responsible nephrologist.
* Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment Target | Baseline
  Feasibility of toolkit will be confirmed if recruitment target of 30 participants at each site are obtained in a 3-month period of the pilot.
Proportion of Eligible Patients who decline consent | Baseline
  Feasibility of toolkit will be confirmed if decline rate is <50% for eligible patients.
Proportion of Participants who miss or refuse ePROMs follow-ups | Baseline to follow-up (6 months)
  Feasibility of toolkit will be confirmed if <30% of participants complete <50% of all follow-up visits.
Proportion of Enrolled Patients who Drop-Out From the Study | Baseline to follow-up (6 months)
  Feasibility of toolkit will be confirmed if the dropout rate is < 30%.

SECONDARY OUTCOMES:
Patient Acceptability | Follow-up (every 4 weeks, up to 6 months)
  Proportion of patients who find the tool 1) acceptable, 2) not burdensome and 3) important, based on responses to the "Patient Satisfaction Survey" they will complete.
Clinical Team Acceptability | Follow-up (every 4 weeks, up to 6 months)
  Proportion of staff who do not find the use of the tool intrusive to the workflow, based on responses to the "Staff Satisfaction Survey" they will complete.

OTHER OUTCOMES:
Incidence Rate of Healthcare Use | Baseline to Follow-up (6 months)
  Patients will complete the 'Healthcare Use Questionnaire' at each follow-up visit. Incidence rate of healthcare use will be determined via incidence of hospitalization and emergency visits every 4 weeks.
Physical Health Component Score | Baseline to Follow-up (6 months)
  Measured by the 36-Item Kidney Disease Quality of Life Instrument (KDQOL-36) and the 12-Item Short Form Health Survey (SF-12) embedded in ePROMs. SF-12 is a part of KDQOL-36, specifically items 1-12. Scoring wise, items 1, 8, & 12-36 have a minimum value of 1 and maximum value of 5. Items 2 & 3 have a minimum value of 1 and maximum value of 3. Items 4-7 have a minimum value of 1 and maximum value of 2. Items 9-11 have a minimum value of 1 and maximum value of 6. Whether higher or lower scores determine better outcomes depends on the item.
Mental Health Component Score | Baseline to Follow-up (6 months)
  Measured by the 36-Item Kidney Disease Quality of Life Instrument (KDQOL-36) and the 12-Item Short Form Health Survey (SF-12) embedded in ePROMs. SF-12 is a part of KDQOL-36, specifically items 1-12. Scoring wise, items 1, 8, & 12-36 have a minimum value of 1 and maximum value of 5. Items 2 & 3 have a minimum value of 1 and maximum value of 3. Items 4-7 have a minimum value of 1 and maximum value of 2. Items 9-11 have a minimum value of 1 and maximum value of 6. Whether higher or lower scores determine better outcomes depends on the item.
Kidney Disease Quality of Life | Baseline to Follow-up (6 months)
  Measured by the 36-Item Kidney Disease Quality of Life Instrument (KDQOL-36). Scoring wise, items 1, 8, & 12-36 have a minimum value of 1 and maximum value of 5. Items 2 & 3 have a minimum value of 1 and maximum value of 3. Items 4-7 have a minimum value of 1 and maximum value of 2. Items 9-11 have a minimum value of 1 and maximum value of 6. Whether higher or lower scores determine better outcomes depends on the item.

CONTACTS AND LOCATIONS:
Overall Officials: Istvan Mucsi, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Etobicoke General Hospital, Brampton, Ontario
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound purpose to achieve aims in the approved proposal or for individual participant data meta-analysis. Proposals should be directed to istvan.mucsi@uhn.ca. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website.

REFERENCES:
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Spitzer RL, Williams JB, Kroenke K, Hornyak R, McMurray J. Validity and utility of the PRIME-MD patient health questionnaire in assessment of 3000 obstetric-gynecologic patients: the PRIME-MD Patient Health Questionnaire Obstetrics-Gynecology Study. Am J Obstet Gynecol. 2000 Sep;183(3):759-69. doi: 10.1067/mob.2000.106580. PMID 10992206
- [Background] Davison SN, Jhangri GS, Johnson JA. Longitudinal validation of a modified Edmonton symptom assessment system (ESAS) in haemodialysis patients. Nephrol Dial Transplant. 2006 Nov;21(11):3189-95. doi: 10.1093/ndt/gfl380. Epub 2006 Sep 6. PMID 16957010
- [Background] Bruce B, Fries JF. The Stanford Health Assessment Questionnaire: dimensions and practical applications. Health Qual Life Outcomes. 2003 Jun 9;1:20. doi: 10.1186/1477-7525-1-20. PMID 12831398
- [Background] Garin O, Ayuso-Mateos JL, Almansa J, Nieto M, Chatterji S, Vilagut G, Alonso J, Cieza A, Svetskova O, Burger H, Racca V, Francescutti C, Vieta E, Kostanjsek N, Raggi A, Leonardi M, Ferrer M; MHADIE consortium. Validation of the "World Health Organization Disability Assessment Schedule, WHODAS-2" in patients with chronic diseases. Health Qual Life Outcomes. 2010 May 19;8:51. doi: 10.1186/1477-7525-8-51. PMID 20482853
- [Background] Van Belle S, Paridaens R, Evers G, Kerger J, Bron D, Foubert J, Ponnet G, Vander Steichel D, Heremans C, Rosillon D. Comparison of proposed diagnostic criteria with FACT-F and VAS for cancer-related fatigue: proposal for use as a screening tool. Support Care Cancer. 2005 Apr;13(4):246-54. doi: 10.1007/s00520-004-0734-y. Epub 2004 Nov 12. PMID 15549424
- [Background] Tam E, Chen J, Zhang Q, et al. Routine physical function assessment through a Branching Logic Electronic Symptom Survey (BLESS) vs. the 32-combined item HAQ-DI + WHODAS (HW) survey: A quality improvement controlled trial. Journal of Clinical Oncology 2017;35:136.
- [Background] Howell D, Liu G. Can routine collection of patient reported outcome data actually improve person-centered health? Healthc Pap. 2011;11(4):42-7; discussion 55-8. doi: 10.12927/hcpap.2012.22703. PMID 22543292
- [Background] Dudgeon D, King S, Howell D, Green E, Gilbert J, Hughes E, Lalonde B, Angus H, Sawka C. Cancer Care Ontario's experience with implementation of routine physical and psychological symptom distress screening. Psychooncology. 2012 Apr;21(4):357-64. doi: 10.1002/pon.1918. Epub 2011 Feb 8. PMID 21308858
- [Background] Barbera L, Sutradhar R, Howell D, Sussman J, Seow H, Dudgeon D, Atzema C, Earle C, Husain A, Liu Y, Krzyzanowska MK. Does routine symptom screening with ESAS decrease ED visits in breast cancer patients undergoing adjuvant chemotherapy? Support Care Cancer. 2015 Oct;23(10):3025-32. doi: 10.1007/s00520-015-2671-3. Epub 2015 Feb 26. PMID 25711657
- [Derived] Gill JK, Pucci M, Samudio A, Ahmed T, Siddiqui R, Edwards N, Marticorena RM, Donnelly S, Lok C, Wentlandt K, Wolofsky K, Mucsi I. Self-reported MeasUrement of Physical and PsychosOcial Symptoms Response Tool (SUPPORT-dialysis): systematic symptom assessment and management in patients on in-centre haemodialysis - a parallel arm, non-randomised feasibility pilot study protocol. BMJ Open. 2024 Jan 30;14(1):e080712. doi: 10.1136/bmjopen-2023-080712. PMID 38296283